CLINICAL TRIAL: NCT02981797
Title: Assess Gamma H2AX Positivity in Circulating Prostate Cancer Cells Before and After Radium 223 Treatment
Brief Title: Assess Gamma H2AX Positivity in Circulating Prostate Cancer Cells Before and After Radium 223
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: MCC-17725; ONC-2013-067 (Other: Bayer Corporation)
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: symptomatic bone metastasis; metastatic; castration resistant
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radium 223 Standard of Care: Standard of Care and Blood Collection for Baseline Circulating Tumor Cells (CTCs) Numeration and H2AX Assay. Participants who have chosen Radium 223 treatment for their prostate cancer that has spread to the bone and causing pain. Week 1 starts with the first Radium 223 treatment and week 24 ends 4 weeks after the last or sixth Radium 223 treatment. The circulating prostate cancer cell analysis will be performed within 24 hours of blood draw. Any unused blood samples for circulating prostate cancer cell analysis will be disposed per lab protocol.
  Interventions: Other: Blood Collection During Standard of Care Treatment

INTERVENTIONS:
Other: Blood Collection During Standard of Care Treatment — Blood collection for baseline CTC numeration and H2AX assay. Circulating prostate cancer cell analysis requires blood draw of 7.5 ml (about 1 ½ teaspoons) of blood, to be performed at the screening, 1-2 hours before the third and sixth dose of radium 223 and 24 hours after the first, third, sixth dose of Radium 223. Standard of care Radium 223 treatment is given every 4 weeks for a total of 6 treatments and post Radium 223 follow up at week 24 is also considered standard of care. Other than these standard clinic visits and treatments, the study only requires 3 extra trips to the cancer center for blood draw at 24 hours after the first, third, sixth dose of Radium 223. Blood draws other than circulating tumor cell analysis is considered standard of care and doesn't require extra visits.

SUMMARY:
This is a prospective biomarker study on prostate cancer patients receiving Radium 223 as standard of care.

Participants will take part in this research study because they have chosen Radium 223 treatment for their prostate cancer that has spread to the bone and causing pain. Investigators want to find out if a blood test performed before and after the Radium 223 treatment will help to understand how prostate cancer cells react to this therapy.

In this pilot study, researchers want to find out if Radium 223 given as part of standard treatment for prostate cancer can decrease the number of circulating prostate cancer cells. Radium 223 kills prostate cancer cells by damaging their DNA. Other than looking at the changes in the number of circulating prostate cancer cells before and after Radium 223, researchers would also like to look at the changes in a DNA damage marker, called gamma H2AX, in the circulating prostate cancer cells before and after treatment with Radium 223. Assessing the DNA damage marker gamma H2AX is investigational. It is performed in the same tube of blood that is used for assessing the changes in the number of circulating prostate cancer cells.

DETAILED DESCRIPTION:
In this pilot study, researchers want to find out if Radium 223 given as part of standard treatment for prostate cancer can decrease the number of circulating prostate cancer cells. Radium 223 kills prostate cancer cells by damaging their DNA. Other than looking at the changes in the number of circulating prostate cancer cells before and after Radium 223, researchers would also like to look at the changes in a DNA damage marker, called gamma H2AX, in the circulating prostate cancer cells before and after treatment with Radium 223. Assessing the DNA damage marker gamma H2AX is investigational. It is performed in the same tube of blood that is used for assessing the changes in the number of circulating prostate cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Male patients 18 years or older
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Receiving radium 223 as standard of care for symptomatic metastatic castration resistant prostate cancer to the bone as documented by bone scan or Sodium Fluoride positron emission tomography (PET) bone scan.
* No evidence of visceral metastasis
* Prior surgical castration or concurrent use of GnRH analogue (i.e., medical castration) with testosterone at screening <50 ng/dL.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 -2, ECOG 3 is allowed if due to pain
* Adequate organ function: Serum alanine aminotransferase (ALT) or aspirate aminotransferase (AST) must be < 2.5 x upper limit of normal (ULN); Total bilirubin < 1.5 s ULN; Estimated creatinine clearance must be >40 mL/min; Absolute neutrophil count (ANC) > 1500/l; Hemoglobin above 10 g/dl; platelet count > 100,000/l.
* Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections or major surgery within 28 days prior to study enrollment
* Life expectancy of 6 months or more
* Must agree to practice effective barrier contraception during the entire study treatment period & through for 6 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse
* Able to give written informed consent
* Have at least 2 CTCs at baseline

Exclusion Criteria:

* Exposure to radioisotope therapy (samarium 153, strontium 89) within 24 weeks or exposure to external beam radiation within 12 weeks of receiving the first dose of Radium 223
* Documented central nervous system metastases, has a history of seizure, stroke or transient ischemic attack (TIA)
* Treatment with any investigational compound within 30 days prior to the first dose of study drugs
* Diagnosis or treatment for another systemic malignancy within 2 years before the first dose of study drugs, or previously diagnosed with another malignancy & have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* New York Association Class III or IV heart failure
* Known human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C, life threatening illness unrelated to cancer, or any serious medical or psychiatric illness that could, in investigators opinion, potentially interfere with participation in this study.
* Potential participants with delayed healing of wounds, ulcers, and/or bone fractures
* Inability to comply with protocol requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have chosen Radium 223 treatment as Standard of Care, for their prostate cancer that has spread to the bone and causing pain.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Changes in Gamma H2AX Positivity | 24 weeks per participant
  Assess changes in gamma H2AX positivity in circulating prostate cancer cells before and after Radium 223 treatment. CTC numeration, the gamma-H2AX detection and interpretation will be performed by Veridex with the cell search platform.
Changes in Circulating Prostate Cancer Cell Numbers | 24 weeks per participant
  Assess changes in circulating prostate cancer cell numbers before and after Radium 223 treatment. CTC numeration, the gamma-H2AX detection and interpretation will be performed by Veridex with the cell search platform.

SECONDARY OUTCOMES:
Pain Response | Up to 24 weeks
  Pain response based on Brief Pain Inventory. Pain will be assessed using the Brief Pain Inventory (BPI) Items #3 (worst pain over the last 24 hours by recall), #5 (average pain over the past 24 hours by recall) and #9 (interference with daily activities and sleep).
Changes in Narcotic Analgesic Use | Up to 24 weeks
  Changes in narcotic analgesic use in participants requiring narcotics at baseline at each radium 223 treatment and week 24. Participants will self-report analgesic use over the past 24 hours.
PSA Response | At week 12
  PSA response (30% decline of pretreatment PSA) at week 12.

OTHER OUTCOMES:
Bone Scan Response | Up to 24 weeks
  Bone scan response based on bone scan index at week 12 and week 24 from dose 1 radium 223 treatment compared with baseline. Response based on the prostate cancer work group 2 (PCWG2) criteria will be assessed at week 12 and week 24 from dose 1 radium 223 treatment and compared with the baseline bone scan.
Changes in Alkaline Phosphatase | Up to 24 weeks
  Changes in alkaline phosphatase at week 12, week 24 compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/